CLINICAL TRIAL: NCT02747849
Title: Pilot Study: Hand & Foot Neuromodulation for Nocturnal Enuresis in Children
Brief Title: Hand & Foot Nocturnal Enuresis TENS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajeev Chaudhry (Other)
Collaborators: The Coulter Foundation (Other)
Responsible Party: Sponsor-Investigator, Rajeev Chaudhry, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro15120157
Record Dates: First submitted 2016-04-05; First posted 2016-04-22 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Bedwetting
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Transcutaneous Electric Nerve Stimulation

ARMS (2):
- Hand neuromodulation (Placebo Comparator): The stimulation characteristics for this arm include a continuous frequency of 5 Hz, pulsewidth 0.2 ms, and intensity 2-4 times the threshold voltage required for finger twitching - or the intensity that the subject feels comfortable with. Subjects will be asked to use the stimulator for a minimum of 60 minutes prior to bedtime for two weeks, or longer if they can tolerate it, have the time, and accurately record the total duration. Stimulation will be performed during the first, second, and third weeks of the study.
  Interventions: Device: TENS
- Foot Neuromodulation (Active Comparator): The stimulation characteristics include a continuous frequency of 5 Hz, pulsewidth 0.2 ms, and intensity 2-4 times the threshold voltage required for inducing toe twitching - or the intensity that the subject feels comfortable with. The subjects will be asked to wear socks on their foot to prevent the electrodes from detachment and to stop the stimulation during walking or in any non-resting situation. Subjects will be asked to use the stimulator for a minimum of 60 minutes prior to bedtime for two weeks, or longer if they can tolerate it, have the time, and accurately record the total duration. Stimulation will be performed during the first, second, and third weeks of the study.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Placebo had stimulator placed on hand. Active comparator had stimulator placed on foot. Amount of time, intensity, threshold voltage, pulsewidth and frequency remained the same for both arms.

SUMMARY:
The investigators believe in order to strengthen the evidence in support of transcutaneous foot stimulation in this population the investigators need to move forward with a randomized comparison study using the TENS device on the hand and foot as a control.

DETAILED DESCRIPTION:
Nocturnal enuresis is a common problem in children which can have a dramatic psychological and social impact on quality of life. Neuromodulation by transcutaneous foot stimulation of peripheral tibial nerve branches has been shown to produce a prolonged inhibition of micturition reflex contractions and significantly increase bladder capacity. The investigators primary goal was to evaluate the effect of foot stimulation on the frequency of nocturnal enuresis episodes in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 5 to 18 years old without any specific neurological disorder or urinary tract infection, clinically diagnosed as having nocturnal enuresis AT LEAST 4 episodes per month by history, nocturnal enuresis is a DSM V diagnosable medical condition
2. Currently having no daytime overactive bladder symptoms, i.e. urinary frequency, urgency, or daytime incontinence
3. Having been assessed for and treated if applicable for behavioral etiologies of nocturnal enuresis - consuming excess fluids or specific bladder irritants
4. Having been assessed for and treated if applicable for constipation

Exclusion Criteria:

1. Children with known neurological disorders which may be contributing to nocturnal enuresis episodes
2. Children found through history to have significant behavioral causes of nocturnal enuresis including consumption of excessive fluids or known bladder irritants
3. Children with chronic constipation who are non-compliant with previous pharmacologic efforts to treat.
4. Children who are not adequately potty trained
5. Children with significant daytime symptoms of overactive bladder including frequency, urgency, and daytime incontinence
6. Children who do not tolerate initial stimulation training session in the urology clinic upon enrollment
7. Children with any implantable medical devices such as a pacemaker will be excluded from the study

Note: Any patient currently taking medication such as an anti-muscarinic or a tricyclic antidepressant for overactive bladder at time of enrollment will be eligible to participate and will be continued on their usual medication and dosage throughout the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Chaudhry, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh og UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hand Neuromodulation | Foot Neuromodulation
Started | 13 | 14
Completed | 12 | 14
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hand Neuromodulation | Foot Neuromodulation | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 14 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [8 to 17] | 12.1 [8 to 17] | 12 [8 to 17]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 9 | 9 | 18
  Gender: Female | 3 | 4 | 7
  Gender: Did not identify | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Nights Wet Per 2 Weeks
Description: The subject/parents will be instructed to record a night-time voiding log specifying the change in number of nights wet per 2 weeks. This log is included in the IRB application. Subjects/parents will fill out the log for a two week period prior to foot stimulation to determine a baseline average of nocturnal enuresis episodes, during week 3 and 4 of the study the subjects will stimulate either their foot or hand to measure any acute effect on nocturnal enuresis episodes and finally during week 5 and 6 of the study, after stimulation subjects will keep a log to evaluate any post-stimulation residual benefit
Time Frame: 6 weeks
Population: Patients with primary nocturnal enuresis.
Measure: Mean (Standard Deviation); unit: # nights wet over 2 weeks
Arm/Group | Hand Neuromodulation | Foot Neuromodulation
Number analyzed (Participants) | 12 | 14
# nights wet over 2 weeks
  # nights wet before stimulation over 2 weeks | 11 (3.46) | 8.78 (4.12)
  # nights wet during stimulation over 2 weeks | 8.75 (3.99) | 6.22 (4.21)
  # nights wet after stimulation over 2 weeks | 9.5 (3.82) | 6.78 (5.19)

2. Primary Outcome: Response to Treatment
Description: Total number of participants that responded to treatment after stimulation with Hand or Foor unit.
Time Frame: An average of 6 weeks
Population: Patients
Measure: Count of Participants; unit: Participants
Groups:
- Hand: Participants that used hand modulation.
- Foot: Participants that used Foot modulation
Arm/Group | Hand | Foot
Number analyzed (Participants) | 12 | 14
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Hand Neuromodulation | Foot Neuromodulation
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT02747849/Prot_SAP_000.pdf